CLINICAL TRIAL: NCT00712452
Title: Evaluation of Chemotherapy Influence on Clinical and Biological Markers of Ovarian Reserve.
Acronym: IROCHIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problems of insuffisant recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: P070707
Record Dates: First submitted 2008-07-02; First posted 2008-07-10 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Infertility
Keywords: fertility; chemotherapy
MeSH Terms: conditions — Infertility | interventions — Biological Factors; Cyclophosphamide; Fluorouracil; Taxoids; Doxorubicin; Vinblastine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): systemic lupus erythematosus
  Interventions: Other: Biology and ultrasonography after chemotherapy
- 2 (Other): breast cancer
  Interventions: Other: Biology and ultrasonography after chemotherapy
- 3 (Other): Hodgkin disease
  Interventions: Other: Biology and ultrasonography after chemotherapy

INTERVENTIONS:
Other: Biology and ultrasonography after chemotherapy — Study of markers of ovarian reserve: Estradiol, LH, FSH and progesterone levels and ultrasonographic antral follicle count (no made in current practice)
  Other Names: cyclophosphamide
  Arms: 1
Other: Biology and ultrasonography after chemotherapy — Study of markers of ovarian reserve: Estradiol, LH, FSH and progesterone levels and ultrasonographic antral follicle count (no made in current practice)
  Other Names: 5FU, épirubicine, cyclephosphamide, taxanes
  Arms: 2
Other: Biology and ultrasonography after chemotherapy — Study of markers of ovarian reserve: Estradiol, LH, FSH and progesterone levels and ultrasonographic antral follicle count (no made in current practice)
  Other Names: adriamycine, bléomycine, vinblastine, daunorubicine
  Arms: 3

SUMMARY:
The objective is to evaluate the influence of chemotherapy, either for auto-immune disease, either for carcinologic disease, on clinical and biological markers of ovarian reserve, for young patients, with normal reproductive functions.

DETAILED DESCRIPTION:
The study will enrol patients between 18 and 35 years, treated with neoadjuvant or adjuvant chemotherapy for systemic lupus erythematosus (Group 1), breast cancer (Group 2) or Hodgkin disease (Group 3)to evaluate the clinical and biological markers of ovarian reserve. The follow-up will last 24 months for each patients with a visit before treatment, and at 3 months, 6 months, one year and two years after treatment.

During this period, we will collect pre and post treatment clinical data,and biological data and ultrasonographic data such as antral follicle count which is a marker of ovarian follicle reserve.These data were not observed in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Women volunteers treated by chemotherapy,
* ≥ 18 and ≤ 35 years old
* Regular menstrual cyclicity, between 25 and 35 days
* Social security affiliation
* Signed informed consent

Exclusion Criteria:

* Women < 18 and > 35 years old
* Pregnancy
* Emergent treatment necessity
* No social security affiliation
* Virgin patients

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AMH level and antral follicle count | one year after the chemotherapy treatment

SECONDARY OUTCOMES:
AMH level and antral follicle count at each visit | 3 months, 6 months, and two years after the chemotherapy treatment
Hormonal status (Estradiol, LH, FSH and progesterone levels) | 3 months, 6 months, and two years after the chemotherapy treatment
Menstrual cyclicity | 3 months, 6 months, and two years after the chemotherapy treatment
pregnancy | 3 months, 6 months, and two years after the chemotherapy treatment
infertility treatment if required | 3 months, 6 months, and two years after the chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Renato Fanchin, MD, Study Director — Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère
Locations (1):
- AP-HP Hôpital Antoine Béclère, Clamart, France